CLINICAL TRIAL: NCT00193440
Title: Phase II Trial of Rituximab and Short Duration Chemotherapy Followed by Zevalin as First-Line Treatment for Patients With Low Grade Follicular Non-Hodgkin's Lymphoma
Brief Title: Rituximab and Chemotherapy Followed by Ibritumomab Tiuxetan as Treatment for Low Grade Follicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Biogen (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LYM 22; 106-PO69
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2010-12

CONDITIONS: Non-Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; ibritumomab tiuxetan

INTERVENTIONS:
Drug: Rituximab
Drug: CHOP
Drug: CVP
Drug: Ibritumomab Tiuxetan

SUMMARY:
In this trial, we will evaluate the feasibility, toxicity, and effectiveness ibritumomab tiuxetan, when incorporated into combination first-line treatment for follicular lymphoma. Addition of the ibritumomab tiuxetan to our previously evaluated, well tolerated combination of rituximab and short course chemotherapy will allow the use of additional active agent with a unique mechanism of cytotoxicity. In addition, "debulking" of lymphoma prior to 90Y Zevalin administration may minimize the myelotoxicity of this agent.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be receive:

* Rituxan + CHOP or CVP + Ibritumomab Tiuxetan

Patients who are considered medical candidates for doxorubicin should receive CHOP chemotherapy (Cyclophosphamide, doxorubicin, vincristine and prednisone). Patients who are not considered medical candidates for doxorubicin should receive CVP chemotherapy (Cyclophosphamide, Vincristine, and prednisone)

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Histologic documentation of follicular center, B-cell lymphoma
* Early stage lymphoma (stages I or II) relapsed after radiation therapy alone
* No previous chemotherapy or monoclonal antibody therapy
* Measurable or evaluable disease
* Able to perform activities of daily living with minimal assistance
* Age > 18 years
* Adequate bone marrow ,liver and kidney function
* Must be accessible for treatment and follow-up.
* Bone marrow examination initial staging and accurate restaging
* All patients must give written informed consent prior to study entry.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Small lymphocytic (CLL type) lymphomas and CLL
* Impaired bone marrow reserve
* Female pregnant or lactating
* Serious active infection at the time of treatment
* Any other serious underlying condition
* Central nervous system involvement (brain or meningeal)
* HIV or AIDS-related lymphoma
* Received prior external beam radiation therapy to > 25% of active bone marrow
* Pleural effusion
* Received prior murine antibodies or proteins
* History of other neoplasms within five years of diagnosis

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-04; Primary Completion 2004-04 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Overall clinical response rate
Overall molecular response rate

SECONDARY OUTCOMES:
Progression-free survival
Overall survival
Overall toxicity

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Hainsworth JD, Spigel DR, Markus TM, Shipley D, Thompson D, Rotman R, Dannaher C, Greco FA. Rituximab plus short-duration chemotherapy followed by Yttrium-90 Ibritumomab tiuxetan as first-line treatment for patients with follicular non-Hodgkin lymphoma: a phase II trial of the Sarah Cannon Oncology Research Consortium. Clin Lymphoma Myeloma. 2009 Jun;9(3):223-8. doi: 10.3816/CLM.2009.n.044. PMID 19525191